CLINICAL TRIAL: NCT03645252
Title: Impact of the Sequence of Vessel Interruption During Major Pulmonary Resections for Non-small Cell Lung Cancer Based on Circulating Tumor Cells Detection Peroperatively in the Tumor-draining Pulmonary Vein: a Randomized Pilot Study.
Brief Title: Sequence of Vessel Interruption and Circulating Tumor Cells in Surgical Lung Cancer
Acronym: CTC-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Collaborators: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Massimo Conti, Medical Doctor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019-2997, 21621
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Circulating Tumor Cell; Lung Cancer; Surgery
MeSH Terms: conditions — Neoplastic Cells, Circulating; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vein first (Active Comparator): Tumor-draining pulmonary vein is interrupted first and before any surgical manipulation.
  Interventions: Procedure: Vein interruption before any other surgical manipulation
- Arteries before vein (Active Comparator): Lobar arteries (+/- bronchus and inter-lobar fissures) are interrupted before tumor-draining pulmonary vein.
  Interventions: Procedure: Arteries interruption before vein interruption

INTERVENTIONS:
Procedure: Vein interruption before any other surgical manipulation — The pulmonary tumor-drainage vein is first exposed and punctured with a 23-gauge needle, and 7.5 ml of blood is drawn from the pulmonary vein prior to subsequent surgical manipulation for lobectomy. Collected blood is versed in a Cellsearch tube provided by the manufacturer (Menarini Silicon Biosystems, Castel Maggiore, Italy).
  In the "vein first" group, the lobar vein is dissected and the cartridge and anvil of a vascular cartridge stapler are placed on either side of the vein. The vein is punctured above the stapler with a 23-gauge needle and 7.5 ml of blood is drawn. Finally, the vein is cut. The intervention then proceeds in the usual manner.
  Arms: Vein first
Procedure: Arteries interruption before vein interruption — The pulmonary tumor-drainage vein is first exposed and punctured with a 23-gauge needle, and 7.5 ml of blood is drawn from the pulmonary vein prior to subsequent surgical manipulation for lobectomy. Collected blood is versed in a Cellsearch tube provided by the manufacturer (Menarini Silicon Biosystems, Castel Maggiore, Italy).
  In the "arteries before vein" group, lobar arteries are first dissected and interrupted (+/- the bronchus and inter-lobar fissures). The lobar vein is then dissected and blood sample is performed as described above.
  Arms: Arteries before vein

SUMMARY:
This study aims to define the impact of the sequence of vessel interruption on change in CTC and CTC clusters density in the tumor-draining pulmonary vein between the period before surgical manipulation and before tumor-draining vein interruption.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC with preoperative pathological evidence,
* Pure solid nodule or part-solid (>50%) ground glass nodule on CT scan
* Clinical stage tumor-1 to 3, clinical stage node-0, clinical stage metastasis-0, (except clinical stage tumor-3 for chest wall, pericardium or phrenic nerve invasion)
* Video-assisted thoracoscopic lobectomy or bi-lobectomy

Exclusion Criteria:

* Pneumonectomy, segmentectomy, non anatomic resection
* History of thoracic surgery on the same side
* Necessity to perform a non-anatomic resection in addition to the lobectomy
* No preoperative histological diagnosis
* Pure ground glass nodule on CT scan
* Clinical stage tumor-4 or 3 for chest wall, pericardium or phrenic nerve invasion
* Clinical stage node ≥1
* Neoadjuvant therapy
* Second cancer or cancer in the past 5 years
* First approach through thoracotomy with ribs spreading
* Pregnancy, <18 years of age
* Pulmonary adherences/symphysis found during surgery (impossible to perform the first blood sample without lung manipulation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-31 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in CTC density | Within 96 hours after surgery
  Changes in CTC count in 7.5 ml of blood sampled from the tumor-draining vein between the period before surgical manipulation (first sample) and before tumor-draining vein interruption (second sample).
Changes in CTC clusters density | Within 96 hours after surgery
  Changes in CTC clusters (or CTC micro-emboli defined as ≥3 contiguous CTC) count in 7.5 ml of blood sampled from the tumor-draining vein between the period before surgical manipulation (first sample) and before tumor-draining vein interruption (second sample).

SECONDARY OUTCOMES:
Disease free survival | 2 years and 5 years after surgery
  Disease free survival 2 years and 5 years after surgery and recurrence site (local or distant metastasis).
Overall survival | 2 years and 5 years after surgery
  Overall survival 2 years and 5 years after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Conti, MD, Principal Investigator — Centre de Recherche IUCPQ - Laval University
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crosbie PA, Shah R, Krysiak P, Zhou C, Morris K, Tugwood J, Booton R, Blackhall F, Dive C. Circulating Tumor Cells Detected in the Tumor-Draining Pulmonary Vein Are Associated with Disease Recurrence after Surgical Resection of NSCLC. J Thorac Oncol. 2016 Oct;11(10):1793-7. doi: 10.1016/j.jtho.2016.06.017. Epub 2016 Jul 25. PMID 27468936
- [Result] Hashimoto M, Tanaka F, Yoneda K, Takuwa T, Matsumoto S, Okumura Y, Kondo N, Tsubota N, Tsujimura T, Tabata C, Nakano T, Hasegawa S. Significant increase in circulating tumour cells in pulmonary venous blood during surgical manipulation in patients with primary lung cancer. Interact Cardiovasc Thorac Surg. 2014 Jun;18(6):775-83. doi: 10.1093/icvts/ivu048. Epub 2014 Mar 11. PMID 24618055